CLINICAL TRIAL: NCT02501967
Title: Care Planning for Older Persons With Multiple Conditions: Encouraging a Tailored Approach (COMET): Stage II
Acronym: COMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1410014812
Record Dates: First submitted 2015-07-08; First posted 2015-07-17 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Polypharmacy
Keywords: multiple chronic conditions
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- COMET (Experimental): The intervention consists of completion of the tool (COMET) by means of a 30 minute telephone interview prior to the primary care visit and provision of the tool's output to the patient and primary care physician. The COMET tool takes information about the patient's medications and chronic conditions from the electronic health record, and then supplements this with information obtained by a telephone interview assessing the patient's cognition, social supports, medication adherence, home medication regimen, medication side effects, and health status. In addition, there is a chart review screen to record renal function, blood pressure, and hemoglobin A1C. All of this information is run through a set of algorithms to identify medication reconciliation errors and potentially inappropriate medications.
  Interventions: Other: COMET
- Usual Care (No Intervention)

INTERVENTIONS:
Other: COMET — The intervention consists of completion of the tool by means of a telephone interview prior to the primary care visit and provision of the tool's output to the patient and PCP.
  Arms: COMET

SUMMARY:
The purpose of the proposed project is to pilot-test in the clinic setting a computer-based clinical decision support system (CDSS) designed to optimize medication prescribing for older persons with multiple chronic conditions and polypharmacy.

ELIGIBILITY:
Inclusion Criteria:

* Veterans age 65 years and older.
* Patients should be diagnosed with diabetes and hypertension and be prescribed five or more medications.
* Patients receiving primary care at the West Haven campus of VA Connecticut Healthcare System.

Exclusion Criteria:

* Unable to manage own medications because of cognitive impairment.
* Medications prescribed by physician outside of the VA.
* Severe vision or hearing impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Patient Assessment of Care for Chronic Conditions (PACIC) | Immediately following the primary care visit at which the patient is enrolled in the study
  A modified version of the Patient Assessment of Care for Chronic Conditions (PACIC) will be used. The original tool is a 20 item instrument (100 points total) designed to assess a patients perception of one's health care (for chronic conditions). A higher score indicates a more favorable rating.

SECONDARY OUTCOMES:
Number of changes made to the medication regimen | 3 Month Follow Up
  A chart review will be completed of the 3 months following the clinic appointment at which the patient is enrolled in the study to document any changes that were made to the medication regimen.
Coding of audiotapes of primary care visit | The primary care visit at which the patient is enrolled in the study
  The Active Patient Participation Coding Scheme (APPC) is a validated instrument to assess indicators and facilitators of patient participation. Audio recordings will also be coded for evidence of providers' partnership building in the form of verbal encouragement to ask questions, express opinions, talk about their feelings, and participate in decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Terri R Fried, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare, West Haven, Connecticut, United States